CLINICAL TRIAL: NCT01063946
Title: A Phase I, Open Label Study Investigating the Disposition of 25 mg/m² [14C]-AVE8062 (1.85 MBq, 50 µCi) Administered at Cycle 1 as a 30-minute Intravenous Infusion to Patients With Advanced Solid Tumors
Brief Title: A Study to Investigate the Disposition of Radio-labeled AVE8062 Compound Administered as a 30-minute IV Infusion to Patients With Advanced Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BEX6587; 2008-007824-24 (EudraCT Number)
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-12

CONDITIONS: Neoplasms, Malignant
MeSH Terms: conditions — Neoplasms | interventions — AC 7700

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [14C]-AVE8062 (Experimental): Single, 30 minute, intravenous infusion of 25 mg/m² of [14C]-AVE8062 containing 1.85 MBq (50µCi) at the first cycle, followed by subsequent administrations with non-radiolabelled AVE8062 in combination with cisplatin every 3 weeks, according to the investigator's judgment.
  Interventions: Drug: Ombrabulin (AVE8062)

INTERVENTIONS:
Drug: Ombrabulin (AVE8062) — Pharmaceutical form:concentrate solution
  Route of administration: intravenous infusion

SUMMARY:
Primary Objectives:

* To determine the excretion balance and systemic exposure of radioactivity after intravenous infusion of [14C]-AVE8062 to humans
* To determine the pharmacokinetics of AVE8062 and RPR258063 and their contribution to overall exposure
* To collect samples to determine the metabolic pathways of AVE8062 and identify the chemical structures of the main metabolites

Secondary Objective:

* To assess the safety profile of the drug

DETAILED DESCRIPTION:
The duration of the study for each patient will include approximately 4 weeks of a screening phase prior to first infusion of study drug, 21-day study treatment cycles and end of treatment visit. The patient can continue treatment until disease progression, unacceptable toxicity, or the patient's refusal of further treatment.

ELIGIBILITY:
Inclusion criteria:

* Patients with advanced neoplastic disease that has become refractory to conventional treatment or for which no standard therapy exists.
* Age = or > 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Adequate hematological, hepatic and renal functions

Exclusion criteria:

* Poor metabolizers for CYP2C19, CYP2C9, CYP2D6 and polymorphic UGTs will be excluded from the study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Percentage of radioactive dose excreted in urine, feces and expired air | 3 weeks (end of cycle 1) or 30 days after the first dose
Concentration-time profiles and pharmacokinetic (PK) parameters of total radioactivity in whole blood and plasma; blood over plasma concentration ratios; Concentration-time profile and PK parameters of AVE8062 and RPR258063 in plasma | 3 weeks (end of cycle 1) or 30 days after the first dose

SECONDARY OUTCOMES:
Safety assessment based on Adverse events reporting, laboratory tests according to the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTC) v3.0 grade scaling | 3 weeks (end of cycle 1) or 30 days after the first dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Brussels, Belgium